CLINICAL TRIAL: NCT03242811
Title: Swedish Age Assessment Study -SAAS Study to Deepen the Knowledge of Magnetic Camera Examinations as a Method for Medical Age Assessment
Brief Title: Swedish Age Assessment Study
Acronym: SAAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berit Larsson (Other)
Collaborators: Blekinge Institute of Technology (Other); Ministry of Health and Social Affairs, Sweden (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Berit Larsson, Unit Manager Karolinska Trial Alliance, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SAAS 20170506
Record Dates: First submitted 2017-07-23; First posted 2017-08-08 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Age Determination by Skeleton
Keywords: Medical age assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Examination by MRI (Experimental): MRI scan of knee, ankle and wrist
  Interventions: Diagnostic Test: MRI scan of knee, ankle and wrist

INTERVENTIONS:
Diagnostic Test: MRI scan of knee, ankle and wrist — At the day of the intervention, the subject is informed about the study by a nurse and provides written informed consent.
  Girls must leave urine tests to rule out pregnancy. The questionnaire for the study is answered by the subject and weight and length are measured. The subject is asked to self-assess his/her puberty.
  After detailed information on how a magnetic camera examination is carried out, an examination of five selected growth zones (knee joint, ankle joint including heel leg and wrist) is performed using 1.5 Tesla magnetic camera with dedicated cartilage sequence.
  Other Names: Self assessment of puberty by Tanner scale; Questionnaire on socioeconomics

SUMMARY:
It is important that asylum seekers should have as accurate age assessment as possible and that children's fundamental rights are met by choosing methods based on best available knowledge. The aim is to provide, on the basis of best available knowledge, suggestions for methods of medical age assessment of whether a person is over or under 18 years of age.

The primary issue is to investigate whether five selected growth zones in knee joint, ankle and wrist individually or in combination can better determine the 18-year limit compared with previous research.

DETAILED DESCRIPTION:
Swedish Age Assessment study is conducted with the aim of

* Deepening the knowledge of age-assessment methodology with magnetic camera examinations among born and registered in Sweden aged 14.0 through 21.5 years
* With a magnetic camera, investigate whether five selected growth zones in the knee joint and ankle joint (distal femur, proximal tibia, distal tibia and calcaneus) and distal radius (wrist) individually or in combination can better determine the 18-year limit compared with previous research
* To investigate how gender and growing environment can affect the end of growth zones

ELIGIBILITY:
Inclusion Criteria:

* Healthy children / young adults without prior illness (such as asthma, growth hormone treatment, prolonged peroral cortisone treatment, cancer treatment, diabetes, rheumatic disease) that may have affected growth can be included in the study.

Exclusion Criteria:

* Children or adolescents with ongoing drug treatment for chronic disease.
* Contraindication against MRI examination
* Pregnancy

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 958 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with correctly classified age (below or above 18 years) when 5 different growth zones in the knee, ankle and wrist are examined by MRI and analysed individually and in combination to determine the maturity. | 1 day
  With 1.5 Tesla magnetic camera with dedicated cartilage sequence, selected growth zones will be investigated: knee joint, ankle joint including heel leg and wrist. The non-dominant body half will be investigated. In order to evaluate the growth zone with the highest precision, we have chosen T2-weighted gradient-recalled echo sequence, called mFFE / MERGE® / MEDIC® by various suppliers. The sequence is used in the clinical practice to assess various types of abnormalities in the cartilage. Two independent and blinded child radiologists shall examine MR images of 5 growth zones of each participant. All sections of each growth zone are to be examined and the cut is selected which shows the highest degree of closing / maturity for grading. Each growth zone will be examined and classified as being mature or non-mature.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Diaz, MD, PhD, Principal Investigator — Karolinska Institutet; Johan Sanmartin Berglund, MD, PhD, Principal Investigator — Blekinge Institute of Technology; Carl-Erik Flodmark, MD, PhD, Study Director — Ministry of Health and Social Affairs, Sweden
Locations (2):
- Sweden (2):
  - Blekinge Institute of Technology, Karlskrona
  - Karolinska Institute, Stockholm

IPD SHARING:
Plan to Share IPD: No